CLINICAL TRIAL: NCT03461744
Title: Diagnostic Scoring for Small Bowel Obstruction
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, MD, PhD, Adj. Prof, Helsinki University Central Hospital
Other Study IDs: SBO-DG
Record Dates: First submitted 2018-02-23; First posted 2018-03-12 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Small Bowel Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is difficult to predict which patients with acute small bowel obstruction require operative intervention and which ones can be handled conservatively. Similarly, strangulation remains difficult decision. The rationale for this observative study is to collect prospective cohort of patients with small bowel obstruction to create scoring system to predict early 1) small bowel obstruction resistant to conservative therapy, 2) strangulation.

ELIGIBILITY:
Inclusion Criteria:

* Computed tomography verified acute small bowel obstruction

Exclusion Criteria:

* < 18 years old
* Pregnant
* Abdominal surgery within 30 days prior recruitment
* Inflammatory bowel disease
* Small bowel tumor causing obstruction
* Peritoneal carcinosis
* Intraluminal obstruction (bile stone, bezoar, etc.)
* Large bowel obstruction
* Small bowel obstruction caused by abdominal wall hernia

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presenting to surgical ER with abdominal complain are screened.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Strangulation | Within hospital stay / 30 days from recruitment
  Number of patients with strangulated bowel (reversible or irreversible ischemic bowel)
Need for surgery due to nonresolving small bowel obstruction | Within hospital stay / 30 days from recruitment
  Number of patients needing surgery due to nonresolving small bowel obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Ville Sallinen, Principal Investigator — Helsinki University Central Hospital
Locations (3):
- Finland (3):
  - Helsinki University Hospital, Jorvi hospital, Espoo
  - Helsinki University Hospital, Meilahti hospital, Helsinki
  - Hyvinkää Hospital, Hyvinkää

IPD SHARING:
Plan to Share IPD: Undecided